CLINICAL TRIAL: NCT03670303
Title: Randomized, Controlled Trial of an Educational Intervention to Promote Spectacle Use Among Secondary School Children in Islamabad, Pakistan
Brief Title: Trial of an Educational Intervention to Promote Spectacle Use Among Secondary School Children in Islamabad, Pakistan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Isra University (Other)
Responsible Party: Principal Investigator, Nusrat Nasim, PHD Scholar, Isra University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIRS-IUISB/1602-PHD-005
Record Dates: First submitted 2018-09-12; First posted 2018-09-13 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Refractive Errors; Visual Impairment
MeSH Terms: conditions — Refractive Errors; Vision Disorders | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Study will involve two groups intervention group and no intervention (control) group. each group will include two boys and two girls schools. Educational intervention will be given to two boys and two girls schools. Remaining two boys and two girls schools will not receive educational intervention. Simultaneous follow-ups will be carried out in two groups to assess compliance towards spectacles use.
Who Masked: Outcomes Assessor
Masking Description: It is limitation of study that at base line data collection and data analysis masking is not possible as investigator has to do herself. Only outcome assessor can be masked to see how many students are using spectacles in intervention group and in control group. he will not be aware about type of groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): This group will include randomly selected two boys and two girls schools. Vision screening and refraction will be carried out at base line.Compliance will be assessed at 6 months follow-up after baseline assessment than educational intervention will be given. Six months after intervention compliance will be assessed again.
  Interventions: Behavioral: Educational intervention
- Control group (No Intervention): This group will also include randomly selected two boys and two girls schools. Vision screening and refraction will be carried out at base line.Compliance towards spectacle use will be assessed at 6 months after baseline assessment. No intervention will be given in this group. Compliance will be assessed again at the same time when assessed in intervention group 6 months after the intervention.

INTERVENTIONS:
Behavioral: Educational intervention — Educational intervention will be given by trained optometrists to participants (requiring spectacles) their parents and teachers. Duration of Intervention will be about one hours and it includes:
  1. Lectures on importance of spectacles use including visual materials such as pictures and videos.
  2. An interactive classroom based demonstration carried out by trained optometrist. Children will be asked to read from blackboard, written to be visible with 6/6 vision, while seated at a distance of 6m. After this children will be given their glasses and asked to read again. The purpose of this demonstration is to make children aware of their poor vision and of the potential impact of corrected VA.
  3. Posters
  4. Brochures
  Arms: Intervention group

SUMMARY:
This study is planned to test an educational intervention promoting the use of spectacles among secondary school children. It is based on the hypothesis that educating teachers, parents and children about the importance of wearing spectacles has the potential to increase spectacle wear among children.Reasons for non-compliance towards spectacle use will be explored and educational intervention will be planned considering these reasons. Educational intervention will increase awareness about the importance of spectacles use and reduce the barriers towards spectacle use.Reducing barriers will increase compliance towards spectacles use which will ultimately prevent the avoidable visual impairment.

DETAILED DESCRIPTION:
Aim of this research is to improve school performance and quality of life of children with refractive errors. Planned research will be carried out in eight (4 girls and 4 boys) Public Sector Secondary Schools of Islamabad and vision of students will be tested with standard snellen chart to recruit 120 boys and 120 girls with refractive errors. Students having vision ≤ 6/12 will receive auto refraction and prescription of spectacles will be given after subjective refraction. primary outcome of purchase of glasses will be asessed at three months after prescribing. Follow up after six months of prescribing spectacles will find out compliance towards spectacles. Non-compliant students will be given a questionnaire to provide the reasons for non-compliance towards spectacles. Focus Group Discussions (FGDs) will be conducted with non-compliant students, their teachers and parents to explore reasons of non compliance.

On the basis of information obtained from FGDs an educational intervention will be planned for students, their parents and teahers to explain importance of spectacles. Through stratified randomization schools will be assigned to intervention and control groups. Four schools including two girls and two boys schools will be assigned to intervention group and four schools (two girls and two boys) will be assigned to control group. Educational intervention will be given to intervention group. Six months after the intervention compliance to spectacle wear will be assessed than pre and post intervention compliance in intervention group and between two groups will be compared to assess effectiveness of intervention.

ELIGIBILITY:
Inclusion Criteria:-

1- Children from 6th to 9th grade (approximate age, 11-16 years) of secondary schools in Islamabad.

Exclusion Criteria:

1. Children from 10th grade which is the final grade of secondary schools.
2. Children with eye disorders other than refractive error.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Purchase of Spectacles | 3 months follow-up after baseline visit.
  Observed wear or possession of purchased glasses.

SECONDARY OUTCOMES:
Wear of spectacles | 6months and one year follow-up after baseline visit.
  Observed wear of spectacles

CONTACTS AND LOCATIONS:
Overall Officials: Shaista Habibullah, PhD, Study Director — Director (Tech)
Locations (8):
- Pakistan (8):
  - Islamabad Model School for Boys G-11/2, Islamabad
  - Islamabad Model School for Boys I-10/2, Islamabad
  - Islamabad Model School for Boys I-8/4, Islamabad
  - Islamabad Model School for Boys I-9/4, Islamabad
  - Islamabad Model School for Girls 1-10/4, Islamabad
  - Islamabad Model School for Girls F-6/1, Islamabad
  - Islamabad Model School for Girls F-7/2, Islamabad
  - Islamabad Model School for Girls G-7/1, Islamabad

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR